CLINICAL TRIAL: NCT07295717
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered ALN-4285 in Adult Healthy Volunteers
Brief Title: A Study to Evaluate ALN-4285 in Adult Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALN-4285-001
Record Dates: First submitted 2025-12-10; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers
Keywords: siRNA; RNAi therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALN-4285 (Experimental): Participants will be administered ALN-4285 subcutaneously (SC)
  Interventions: Drug: ALN-4285
- Placebo (Placebo Comparator): Participants will be administered placebo SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALN-4285 — ALN-4285 will be administered SC
  Arms: ALN-4285
Drug: Placebo — Placebo will be administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to:

* evaluate the safety and tolerability of single ascending doses of ALN-4285 in healthy volunteers
* characterize the single-dose pharmacokinetics (PK) of ALN-4285

ELIGIBILITY:
Inclusion Criteria:

* Has a body mass index (BMI) of ≥18.0 kg/m^2 and ≤30 kg/m^2
* Has 12-lead ECG within normal limits or with no clinically significant abnormalities in the opinion of the Investigator

Exclusion Criteria:

* Has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >upper limit of normal (ULN)
* Has total bilirubin >ULN
* Has systolic blood pressure >140 mmHg and/or a diastolic blood pressure >90 mmHg
* Has an estimated glomerular filtration (eGFR) of <90 mL/min/1.73m^2 at screening
* Has received an investigational agent within the last 30 days or 5 half-lives

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-12-12 (Estimated); Primary Completion 2026-12-29 (Estimated); Study Completion 2027-03-23 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events (AEs) | Up to Week 24

SECONDARY OUTCOMES:
Concentration of ALN-4285 in Plasma | Up to Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals Inc
Locations (1):
- Clinical Trial Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No